CLINICAL TRIAL: NCT04118309
Title: The Effects of High-intensity Interval Training on Mental Health and Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Natural Sciences and Engineering Research Council, Canada (Other)
Responsible Party: Principal Investigator, Jennifer Heisz, Associate Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-508
Record Dates: First submitted 2019-10-03; First posted 2019-10-08 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Anxiety; Depressive Symptoms; Inflammation
MeSH Terms: conditions — Anxiety Disorders; Depression; Inflammation | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-intensity interval training (Experimental): Three sessions of high-intensity interval training per week for nine weeks. Following a three minute warm up, a session contained twenty minutes of alternating between a sprint (80% of maximum workload, 90-95% of maximum heart rate) and active rest (30% of maximum workload) at a one minute to one minute ratio. Every session ended with a two and a half minute cool down.
  Interventions: Behavioral: Exercise
- Placebo exercise group (Placebo Comparator): No changes in physical activity behaviour occurred (already engaging in less than 150 minutes per week, instructed to maintain their current inactivity). They were told they needed to stay inactive since they were part of an 'acute' exercise group, aiming to see how long the effects of their baseline maximal exercise test would last. Thus, the cover story gave them the impression they were also in an exercise group, as oppose to a non-exercise control group.
  Interventions: Other: Placebo

INTERVENTIONS:
Behavioral: Exercise
  Arms: High-intensity interval training
Other: Placebo
  Arms: Placebo exercise group

SUMMARY:
The present study investigated the effects of high-intensity interval exercise training and placebo-exercise on mental health and inflammation using a randomized control trial. The study also examined how anxiety symptoms prior to high-intensity interval training may influence improvements in fitness. Inactive young adults underwent nine weeks of either high-intensity interval training or their regular routine. Questionnaires, a blood draw and a maximal exercise test were conducted the week before and week after the intervention. It was hypothesized those who underwent high-intensity interval training would experience greater reductions in their depression, anxiety, and inflammation than those who were in the placebo control group. It was also hypothesized those who had high anxiety symptoms at the start of high-intensity interval training would experience smaller improvements in fitness than those who had low anxiety symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Full-time student at McMaster University
* Speak, read and understand English

Exclusion Criteria:

* Exercising for more than 150 minutes of moderate-to-vigorous physical activity per week

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-09-14 (Actual); Primary Completion 2016-04-08 (Actual); Study Completion 2016-04-08 (Actual)

PRIMARY OUTCOMES:
Change in mental illness symptoms (anxiety, depression) from baseline to post-intervention | 11 weeks
  The 21-items of the Beck Anxiety Inventory (Beck, Brown, Epstein & Steer, 1998) are summed to produce a total score from 0-63, with a higher score reflecting more severe anxiety symptoms. The 21-items of the Beck Depression Inventory (Beck, Steer, & Brown, 1996) are summed to produce a total score from 0-63, with a higher score reflecting more severe depressive symptoms.
Change in concentration of circulating proinflammatory cytokines (Interleukin-6, Interleukin-1 beta, Tumour necrosis factor alpha) from baseline to post-intervention | 11 weeks
  Picogram measured from venous blood sample
Change in cardiorespiratory fitness from baseline to post-intervention | 11 weeks
  VO2peak test (ml/min/kg)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Heisz, PhD, Principal Investigator — McMaster University

IPD SHARING:
Plan to Share IPD: No
The sharing of individual data with other researchers was not included in the informed consent signed by participants. Therefore, individual data will not be released.

REFERENCES:
- [Background] Paolucci EM, Loukov D, Bowdish DME, Heisz JJ. Exercise reduces depression and inflammation but intensity matters. Biol Psychol. 2018 Mar;133:79-84. doi: 10.1016/j.biopsycho.2018.01.015. Epub 2018 Feb 3. PMID 29408464
- [Background] Reiss S, Peterson RA, Gursky DM, McNally RJ. Anxiety sensitivity, anxiety frequency and the prediction of fearfulness. Behav Res Ther. 1986;24(1):1-8. doi: 10.1016/0005-7967(86)90143-9. No abstract available. PMID 3947307
- [Background] Stubbs B, Rosenbaum S, Vancampfort D, Ward PB, Schuch FB. Exercise improves cardiorespiratory fitness in people with depression: A meta-analysis of randomized control trials. J Affect Disord. 2016 Jan 15;190:249-253. doi: 10.1016/j.jad.2015.10.010. Epub 2015 Oct 23. PMID 26523669